CLINICAL TRIAL: NCT00304902
Title: Retrospective Chart Review of the Outcome of Treatment for Staphylococcus Aureus Bacteremia
Brief Title: Chart Review of Outcome of Treatment for S. Aureus Bacteremia
Status: Completed | Type: Observational
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Nancy Logan, MA, VAMC
Other Study IDs: H-18867
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-09

CONDITIONS: Staphylococcus Aureus
Keywords: MRSA; Methicillin Resistant Staphylococcus aureus; Staphylococcus aureus Bacteremia
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to review medical records at MEDVAMC in order to relate the outcome of bacteremic MRSA infection to the antibiotics selected for treatment.

DETAILED DESCRIPTION:
Treatment of bacteremic infection (infection associated with positive blood cultures) due to Staphylococcus aureus has become increasingly problematic as a result of the increasing prevalence of strains that are resistant to beta-lactam antibiotics (so-called methicillin-resistant Staphylococcus aureus, MRSA). About 70% of hospital-related strains of S. aureus are MRSA, and, in the past 4 years, the incidence of MRSA in community-acquired infection has risen to about 50%; these data are quite representative of what is being seen elsewhere in the United States and other parts of the world.

Bacteremic MRSA infections are highly problematic for at least two reasons: (1)they are serious, with substantial morbidity and about a 25% rate of mortality in middle-aged adults, the principal patients in our system; and (2)available antibiotic therapy is suboptimal.

In the pre-MRSA era (before 1982 in the United States), treatment of bacteremic S. aureus infection with a beta-lactam antibiotic such as nafcillin produced a uniform microbiological cure (Musher DM, McKenzie SO: Infections due to Staphylococcus aureus. Medicine 56:383-409, 1977). This means that, in the absence of an untreated focus of infection that required surgical removal (such as a myocardial abscess), antibiotics rapidly sterilized the blood stream. This does not mean that no one died; deaths from complications of infection remained common. But, at autopsy, there was generally no evidence for active infection. Extensive literature examined the question of whether gentamicin should be added to nafcillin to treat this kind of disease (reviewed critically in DM, Verner EF: Treatment of Infections due to Staphylococcus aureus. IN The Staphylococci, Ed. by J Jeljascewicz, Gustave Fischer Verlag, Stuttgart, New York, pp.407-419, 1986). Gentamicin produced a synergistic bactericidal effect agains S. aureus in vitro and in animal models. In humans, the addition of gentamicin was associated with more rapid sterilization of the blood stream, but prolonged gentamicin therapy was also associated with nephrotoxicity.

In contrast, in the MRSA era, treatment with vancomycin is associated with persistence of bacteremia (positive blood cultures) and death from active infection. The investigators have recently participated in a prospective observational study that documented the association between vancomycin treatment, persistently positive blood cultures, and persistence of active infection during treatment of S. aureus bacteremia with vancomycin (Chang F-Y, McDonald BB, Peacock, Jr. JE, Musher DM, et al. Staphylococcus aureus bacteremia: recurrence and the impact of antibiotic treatment in a prospective multicenter study. Medicine 82:333-339, 2003).

There appears to be a very close correlation between the outcome of treatment for serious S. aureus infection and the bactericidal activity of the treating antibiotic in vitro using conventional techniques (Musher DM, Verner EF: Treatment of infections due to Staphylococcus aureus. IN The Staphylococci, Ed. by J Jeljascewicz, Gustave Fischer Verlag, Stuttgart, New York, pp.407-419, 1986). We recently showed that adding low concentrations of gentamicin to vancomycin led to substantial synergistic bactericidal activity against MRSA (Shelburne SA, Musher DM, Hulten K, Ceasar H, Lu MY, Bhaila I, Hamill RJ. In-vitro killing of community-associated methicillin-resistant Staphylococcus aureus with drug combinations. Antimicrob Agents Chemother 48:4016-9, 2004).

Based in part on the analogy of nafcillin for treating methicillin-susceptible S. aureus infection, and in part of in vitro studies such as ours (cited above), some physicians regularly add gentamicin to vancomycin for treating MRSA infection. Others, without even the in vitro support, add rifampin either instead of gentamicin or together with gentamicin. There are no clinical studies to support or to refute any of these clinically motivated usages.

Thus, at present, about one-third of patients with MRSA bacteremia at VAMC are treated with vacomycin plus gentamicin, and two-thirds receive vancomycin alone; some in each group receive rifampin. The decisionto add gentamicin is made a haphazard fashion, generally reflecting the interpretation of the literature by the attending physician and/or the residents.

Our proposal is, simply to systematically review records from the past two years in order to relate treatment of MRSA bacteremic infection to outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Staphylococcus aureus in a blood culture between January 1, 2004 and December 31, 2005.

Exclusion Criteria:

* None

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients with Staphylococcus aureus in a blood culture.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2006-02; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Musher, M.D., Principal Investigator — Baylor College of Medicine, Houston VA Medical Center
Locations (1):
- Michael E. DeBakey Veterans Affairs Medical Center, Houston, Texas, United States